CLINICAL TRIAL: NCT01450644
Title: A Fast-track Randomised Controlled Trial to Evaluate a Hospital2Home Palliative Care Service for Patients With Advanced Progressive Idiopathic Fibrotic Interstitial Lung Disease
Brief Title: Evaluation of the Hospital2Home Palliative Care Service for Patients With Advanced Progressive Lung Disease
Acronym: H2H-ILD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCR3669
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Lung Disease
Keywords: Advanced; Progressive; Idiopathic Fibrotic Interstitial Lung Disease; Palliative Care; Randomised; Controlled
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fast track (Other): If patients are randomised to fast-track, their information will be passed to the H2H nurse to organise a case conference within one week of discharge.
  Interventions: Other: The Hospital2Home Service
- Waiting list (Other): If patients are in the control arm, they will continue to receive Standard Best Practice (SBP) and their data will be held by the researcher until after the second interview (4 weeks). After this time, they will be contacted by the H2H nurse to receive the intervention and will be interviewed and followed up as for the fast track group.
  Interventions: Other: The Hospital2Home Service

INTERVENTIONS:
Other: The Hospital2Home Service — This intervention is a new multiprofessional, patient case conference that is organised for people nearing the end-of-life. Evidenced based guidelines for the management of the physical, psychological, spiritual and end of life-planning needs for these patients will be used in the H2H case conference. A case conference will be organised in their home (or place of their choice). The patient, informal caregiver, H2H CNS, GP, district nurse, social worker and community palliative care nurse are invited to attend. Current and anticipated care needs are discussed, and an action plan is agreed allocating a responsible health care professional for each item. During the case conference, individualised care plans will be made. This is then communicated with local services, primary and specialist teams resulting in streamlining of transfer of data and codifying responsibility for the patient, hospital and community care professionals.

SUMMARY:
The investigators hypothesise that H2H will result in improved symptom control and quality of life and may be more cost-effective than standard best practice.

Interstitial Lung Disease (ILD) is a lung condition characterised by progressive scarring - known as fibrosis. This is especially seen in patients with idiopathic pulmonary fibrosis (IPF). There around 2,000 new patients diagnosed in the UK every year with a similar number of deaths.

Fibrotic-ILD causes breathing to slowly deteriorate and as there is no cure, an estimated two-thirds of patients die within five years of diagnosis. Patients suffer from many symptoms including shortness of breath, cough, low mood and fatigue which are currently being poorly managed. In addition, these patients suffer a poor health related quality of life whilst dying from their disease.

In the later stages of their disease, these patients often end up in hospital (see appendix 1a) when there is no proven or effective treatment. Many die there despite wishing to be looked after and die at home. These patients rarely receive palliative care which may help to improve their symptoms, quality of life, address end of life planning needs and prevent hospital admission. The Hospital2Home case conference conducted in the patient's home (or place of their choice) aims to address this. At the case conference involving the patient, their carers, a specialist nurse, and all the community health professionals, a care plan specific to the patient will be developed. Each health professional will be aware of their responsibility and duties. The investigators will look at whether this results in better symptom control and better quality of life for the patient and their carer. The investigators will also examine whether this prevents emergency hospital admission and allows patients to die in their preferred place. The investigators will compare patients who receive the service immediately with those who receive it after a delay.

ELIGIBILITY:
Inclusion Criteria:

Patients i)Clinical diagnosis of PIF-ILD and a 30% survival at 1 year according to the validated prognostic tool developed by Professor Wells.(Appendix 5)

ii) Aged 18 years or over

iii) Any patient who does not meet any of the exclusion criteria

Carers i) The informal caregivers of patients specified above, who can be significant others, relatives, friends or neighbours

ii) Aged 18 years or over

iii) Any carer who does not meet the exclusion criteria

Health professional Primary health professional in contact with patient able to give consent

Exclusion Criteria:

Patients/informal caregiver i) Any patient/ informal caregiver unable to give informed consent

ii) Any patient/informal caregiver less than 18 years of age

iii) Participants who are unable to understand/speak English

iv) Participants who are remaining as an inpatient in the hospital or being transferred to another inpatient facility (eg hospice unit, for terminal care)

v) Participants whose prognosis is less than 1 week or judged too unwell by the research team to take part in serial interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Change in POS scores from week 4 to baseline for each group | 15 months
  POS scores evaluate symptoms and palliative concerns using the Palliative Care Outcome Scale (POS). This comprises eight questions on anxiety, patient and informal caregiver concerns, and practical needs, each rated 0-4. This scoring system will ensure that there is some ongoing data available if the patient becomes unwell and is no longer able to complete the study.

SECONDARY OUTCOMES:
comparison of the patient and informal caregiver POS in this study to see how inter-changeable/reliable the 2 assessments are | 15 months
  At each interview, service use questions will be asked which will record the frequency and types of health/social services received in order that an accurate evaluation of cost of care per patient can be made. In addition semi-structured qualitative interviews will be conducted with patients, informal caregivers and health professionals. Prompts will include views of the case conference, the guidelines and what level of input was needed after the case conference. A record will be made of when and where the patient dies.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Julia Riley, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust, London, London
  - The Royal Brompton NHS Foundation Trust, London, London

REFERENCES:
- [Derived] Bajwah S, Ross JR, Wells AU, Mohammed K, Oyebode C, Birring SS, Patel AS, Koffman J, Higginson IJ, Riley J. Palliative care for patients with advanced fibrotic lung disease: a randomised controlled phase II and feasibility trial of a community case conference intervention. Thorax. 2015 Sep;70(9):830-9. doi: 10.1136/thoraxjnl-2014-206583. Epub 2015 Jun 23. PMID 26103995